CLINICAL TRIAL: NCT05672537
Title: Duvalumab Combined With GemCis Neoadjuvant Therapy of Resectable Intrahepatic Cholangiocarcinoma With High Recurrence Risk, Phase II, Single Center, Randomized Controlled Study
Brief Title: Durvalumab Combined With GemCis Neoadjuvant Therapy of Resectable Intrahepatic Cholangiocarcinoma With High Recurrence Risk
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D20230101
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Durvalumab; Intrahepatic Cholangiocarcinoma; Gemcis
MeSH Terms: conditions — Cholangiocarcinoma | interventions — durvalumab; Surgical Procedures, Operative; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab Combined with GemCis Neoadjuvant Therapy Group (Experimental)
  Interventions: Drug: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin
- Surgical treatment group (Experimental)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Durvalumab — 1500mg intravenous injection for 21d cycle
  Arms: Durvalumab Combined with GemCis Neoadjuvant Therapy Group
Procedure: Surgery — Surgery
  Arms: Surgical treatment group
Drug: Gemcitabine — gemcitabine 1000mg/m2, D1&D8, 21d cycle.
  Arms: Durvalumab Combined with GemCis Neoadjuvant Therapy Group
Drug: Cisplatin — cisplatin 25mg/m2, D1&D8, 21d cycle.
  Arms: Durvalumab Combined with GemCis Neoadjuvant Therapy Group

SUMMARY:
This study is a randomized controlled study to evaluate the efficacy and safety of Durvalumab combined with GemCis for neoadjuvant treatment of high recurrence risk ICC

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, male or female;
2. Pathological diagnosis confirmed intrahepatic cholangiocarcinoma, which could be resected surgically; One of the following conditions shall be met:

   2.1 Single tumor, diameter greater than 5cm (T1b) 2.2 Single tumor with vascular invasion (T2), multiple tumors ≤ 3 2.3 Tumor penetrating visceral peritoneum (T3) or directly invading surrounding organs (T4) 2.4 Suspicious lymph node metastasis in Zone 8, 12 or 13
3. Can not received systemic treatment before participating in the study;
4. ECOG PS score 0-1;
5. The main organs function normally, and there is no serious blood, heart, lung, liver, kidney, bone marrow and other functional abnormalities and immune deficiency diseases.
6. Laboratory inspection shall meet the following requirements:

   Women of childbearing age must have a negative pregnancy test (serum or urine) within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug; For men, they should be surgically sterilized or agree to use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug.
7. The patient voluntarily participated and signed the informed consent form;
8. It is expected that the compliance is good, and the efficacy and adverse reactions can be followed up according to the requirements of the scheme.

Exclusion Criteria:

1. Patients who received PD-1, PD-L1, PD-L2, CTLA-4 before enrollment, or directly received another stimulatory or co inhibitory T cell receptor (such as CTLA-4, 0X40, CD137);
2. Any other research drugs within 4 weeks before enrollment;
3. Any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism after hormone replacement therapy);
4. Congenital or acquired immune function defects, such as human immunodeficiency virus (HIV) infection;
5. Uncontrollable clinical cardiac symptoms or diseases, such as NYHA II and above heart failure unstable angina pectoris, myocardial infarction within one year, and clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
6. Severe infection (such as intravenous drip of antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first drug administration, or fever of unknown cause>38.5 ° C occurred during screening/before the first drug administration;
7. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
8. Live attenuated vaccine shall be inoculated within 4 weeks before the first administration or planned during the study period;
9. Suffered from or accompanied by other system malignant tumors in the last 5 years (except cured skin basal cell carcinoma, cervical carcinoma in situ and ovarian cancer);
10. Allergic to any test drug;
11. Pregnant and lactating women, fertile subjects are unwilling to take effective contraceptive measures;
12. Uncontrollable psychosis;
13. Other situations that the researcher thinks are not suitable for inclusion. If the patient has central nervous system metastasis, has serious laboratory examination abnormalities, and is accompanied by family or social factors, it will affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year relapse free survival rate | 1-year

SECONDARY OUTCOMES:
2-year relapse free survival rate | 2-year
ORR | 1-year
DCR | 1-year
R0 resection rate | 1-year
30 day postoperative complication rate | 30 day
Occurrence of adverse reactions | 1-year
1-year OS | 1-year
2-year OS | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China